CLINICAL TRIAL: NCT01053130
Title: The Effect of Weight Loss Surgery on Preservation of Kidney Function and Cardiovascular Disease Risk Factors in Obese Patients With Stages 3-4 Chronic Kidney Disease: a Randomised Controlled Trial
Brief Title: Weight Loss Interventions in Obese Patients With Stages 3-4 Chronic Kidney Disease: a Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Miss Helen MacLaughlin, King's College Hospital NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCH1639; 09/H0806/69 (Other: UK Research Ethics Committee registration)
Record Dates: First submitted 2010-01-20; First posted 2010-01-21 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2010-01

CONDITIONS: Chronic Kidney Disease; Obesity
Keywords: obesity; bariatric surgery; chronic kidney disease; weight loss; exercise
MeSH Terms: conditions — Renal Insufficiency, Chronic; Obesity; Weight Loss; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- weight loss surgery (Experimental): laparoscopic sleeve gastrectomy
  Interventions: Procedure: laparoscopic sleeve gastrectomy
- Lifestyle Intervention (Active Comparator): Diet and exercise with or without pharmacotherapy
  Interventions: Behavioral: weight management program

INTERVENTIONS:
Procedure: laparoscopic sleeve gastrectomy — laparoscopic sleeve gastrectomy plus dietary and physical activity support
  Arms: weight loss surgery
Behavioral: weight management program — 1200-1500 kcal renal diet, increased physical activity, with optional orlistat therapy at 120 mg tds for 12 months
  Arms: Lifestyle Intervention

SUMMARY:
Weight loss surgery is the most effective weight loss treatment available, but the direct effect on chronic kidney disease is less widely understood. Early research shows some improvement in kidney function may occur and candidacy for kidney transplantation can be improved with weight loss following surgery. To date, no randomised controlled trial has been performed to examine the effect of weight loss surgery on the progression of chronic kidney disease.

This randomised trial will allocate patients to either lifestyle modification with diet, exercise and pharmacotherapy, or weight loss surgery to remove two thirds of the stomach using the laparoscopic sleeve gastrectomy procedure. This study aims to evaluate weight loss surgery vs lifestyle modification in patients with chronic kidney disease with estimated kidney function of 20-60% and morbid obesity (BMI 35-45) in terms of kidney function, cardiovascular disease risk factors and all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

* Stages 3-4 CKD patients (GFR 20-60 mL/min)
* Male or female
* BMI 35-45 kg/m2
* Aged >18 years
* Previously attempted weight loss
* Fit or anesthesia and surgery
* Written informed consent

Exclusion Criteria:

* Pregnancy
* History of chronic liver disease
* Previous gastric surgery or large hiatus hernia
* Previous bariatric surgery
* Psychiatric illness, including anxiety, mood and untreated eating disorders
* Malnutrition (assessed by subjective global assessment)
* Infection or course of antibiotics within the last month
* Unwilling to consider surgical treatment
* Previous kidney transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Measured glomerular filtration rate (renal function) using the iohexol clearance method in patients with stages 3-4 chronic kidney disease | 0, 6, 12 months

SECONDARY OUTCOMES:
Composite end point of death and cardiovascular outcomes (stroke, myocardial infarction or congestive heart failure hospitalisation) | 0, 6, 12, 24, 36 months
Quality of life and anxiety and depression assessment | 0, 6, 12, 24, 36 months
Urinary albumin to creatinine ratio and protein to creatinine ratio | 0, 6, 12, 24, 36 months
Body composition (weight, BMI, waist and hip circ, BIA) | 0, 6, 12 months
Insulin resistance (HOMA method) | 0, 6, 12 months
Serum adiponectin, leptin, IL-6, TNF-α, hs-CRP, fetuin a | 0, 6, 12 months
Urinary markers IL-6, MCP-1, IL-1β, RBP, NAG | 0, 6, 12 months
Endothelial function (flow mediated dilatation) | 0, 6, 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital, London, United Kingdom

REFERENCES:
- [Derived] Conley MM, McFarlane CM, Johnson DW, Kelly JT, Campbell KL, MacLaughlin HL. Interventions for weight loss in people with chronic kidney disease who are overweight or obese. Cochrane Database Syst Rev. 2021 Mar 30;3(3):CD013119. doi: 10.1002/14651858.CD013119.pub2. PMID 33782940